CLINICAL TRIAL: NCT00637728
Title: A Randomized, Double-blind, Placebo-controlled Study of Megestrol Acetate Concentrated Suspension for the Treatment of Cancer-associated Anorexia in Subjects With Lung or Pancreatic Cancer
Brief Title: Treatment of Cancer-anorexia Using Megestrol Acetate Concentrated Suspension in Lung or Pancreatic Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty finding the required patient population
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100.2.C.006 TRANSFERRED
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Anorexia; Cachexia; Weight Loss
Keywords: Megestrol acetate; Anorexia; Cachexia; Lung cancer; Pancreatic cancer; Unintended weight loss; Body weight; Appetite; Megace ES
MeSH Terms: conditions — Anorexia; Cachexia; Weight Loss; Lung Neoplasms; Pancreatic Neoplasms; Body Weight | interventions — Megestrol Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Megestrol acetate concentrated suspension 110 mg/mL
  Interventions: Drug: Megestrol acetate concentrated suspension 110 mg/mL
- 2 (Placebo Comparator): Placebo suspension
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Megestrol acetate concentrated suspension 110 mg/mL — Megestrol acetate concentrated suspension 110 mg/mL given as an oral dose of 550 mg (5 mL) once per day for 56 days, with an optional 28 days extension phase
  Other Names: Megace ES
  Arms: 1
Drug: Placebo — Placebo oral suspension, 5 mL once daily
  Arms: 2

SUMMARY:
Purpose of the study is to compare the effects of megestrol acetate concentrated suspension and placebo on caloric intake for the treatment of cancer-associated anorexia in patients with lung or pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

* Stage II, III,or IV lung or pancreatic cancer
* Fair, poor, or very poor appetite
* Cancer associated anorexia/cachexia
* Weight loss perceived to be associated with diminished appetite
* Eastern Cooperative Oncology Group Performance score of 0, 1, 2
* Life expectancy >3 months
* Alert and mentally competent
* Women of child-bearing potential required to use an adequate and reliable method of contraception. Post-menopausal women have to have been so for at least 1 year
* Screening laboratory values must not be clinically significant (some exceptions per protocol)

Exclusion Criteria:

* Brain, or head and neck metastases that may interfere with food consumption
* AIDS-related wasting
* Radiation therapy to the head and neck, abdomen, or pelvis within past 6 weeks, or anticipated during course of the study such that the result may interfere with food consumption
* Conditions that interfere with oral intake, or ability to swallow
* Absence of a normally functioning gut
* Mechanical obstruction of the alimentary or biliary tract, or malabsorption syndrome
* Intractable or frequent vomiting that regularly interfere with eating
* Clinically significant diarrhea
* History of recurrent thromboembolic events, a thromboembolic event in past 3 months, or long-term anticoagulation treatment for thromboembolism
* Uncontrolled diabetes mellitus, or symptomatic hypoadrenalism
* Poorly controlled hypertension, or congestive heart failure
* Pregnant/lactating females
* Use within past 30 days of an appetite stimulant
* Use within past week, or planned use during the study of parenteral nutrition or tube feedings
* Chronic use of steroids within past 3 months (intermittent short-term use allowed)
* Current use of or not willing to abstain from using illicit substances
* Allergy, hypersensitivity, or contraindication to megestrol acetate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn D Kramer, MD, Study Chair — Par Pharmaceutical, Inc.; John N Mehanna, MD, Principal Investigator — Western Maryland Health System; M.Daud Nawabi, MD, Principal Investigator — Lowcountry Hematology & Oncology, PA; Marc A Saltzman, MD, Principal Investigator — Innovative Medical Research of South Florida, Inc
Locations (3):
- United States (3):
  - Innovative Medical Research of South Florida, Inc, Miami, Florida
  - Western Maryland Health System, Cumberland, Maryland
  - Lowcountry Hematology & Oncology, PA, Mt. Pleasant, South Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After screening, eligible subjects were randomized to treatment in the double-blind phase. After completing the double-blind phase or discontinuing due to specific weight loss criteria, eligible subjects could enter an open-label extension phase.
Groups:
- DB MA-CS 550 mg/Day: Megestrol acetate concentrated suspension (MA-CS; 110 mg/mL) administered orally once every 24 hours (q24h), for a daily dose of 550 mg per day (5 mL dose) in the 8-week double-blind (DB) phase
- DB Placebo: Placebo suspension administered orally q24h (5 mL dose) in the 8-week DB phase
- OL MA-CS 550 mg/Day: MA-CS (110 mg/mL) administered orally q24h, for a daily dose of 550 mg per day (5 mL dose) in the 4-week open-label (OL) extension phase
Period: Double-blind Phase
Arm/Group | DB MA-CS 550 mg/Day | DB Placebo | OL MA-CS 550 mg/Day
Started | 4 | 1 | 0
Completed | 0 | 0 | 0
Not Completed | 4 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Non-compliance | 2 | 0 | 0
Not completed — Study Discontinued | 1 | 1 | 0
Period: Extension Phase
Arm/Group | DB MA-CS 550 mg/Day | DB Placebo | OL MA-CS 550 mg/Day
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received at least 1 dose of study medication and who had at least 1 on-therapy safety assessment
Groups:
- DB MA-CS 550 mg/Day: MA-CS (110 mg/mL) administered orally q24h, for a daily dose of 550 mg per day (5 mL dose) in the 8-week DB phase
- Total: Total of all reporting groups
Arm/Group | DB MA-CS 550 mg/Day | DB Placebo | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Caloric Intake Over the Course of the 8-week Double-blind Phase
Description: The Nutrition Data System for Research (NDSR) was used to determine nutrient and caloric value for foods and beverages consumed and recorded by subjects over a 3-day assessment period prior to each visit. Total number of calories consumed during each 3-day assessment was averaged over available values to determine the week's daily caloric intake value.
Time Frame: 8 weeks
Population: Results not analyzed due to early termination of the study. Study was terminated early, no data were collected for this Outcome Measure.
Arm/Group | DB MA-CS 550 mg/Day | DB Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Changes in Body Composition as Measured by Bioelectric Impedance Analysis (BIA) at Week 4 and Week 8 Relative to Baseline
Time Frame: Baseline, Week 4 and Week 8
Population: as for outcome 1
Arm/Group | DB MA-CS 550 mg/Day | DB Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Weight Over the Course of the 8-week Double-blind Phase
Time Frame: Baseline, Week 1, 2, 3, 4, 6, and 8
Population: as for outcome 1
Arm/Group | DB MA-CS 550 mg/Day | DB Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Appetite Over the 8-week Double-blind Phase as Measured by a VAS Appetite Scale
Description: Subjects marked 6 items on a visual analog scale (VAS) appetite scale including feeling not hungry to hungry, not nauseated to nauseated, empty to full, not satiated to satiated; weak to strong desire to eat; and ability to eat none to a large amount of food
Time Frame: Baseline, Weeks 1, 2, 3, 4, 6 and 8
Population: as for outcome 1
Arm/Group | DB MA-CS 550 mg/Day | DB Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 98 days (from informed consent through 7 days following the last dose of study drug or up until the last protocol-specified study visit, whichever occurred later)
Groups:
- OL MA-CS 550 mg/Day: MA-CS (110 mg/mL) administered orally q24h, for a daily dose of 550 mg per day (5 mL dose) in the 4-week OL extension phase
Arm/Group | DB MA-CS 550 mg/Day | DB Placebo | OL MA-CS 550 mg/Day
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 3/4 | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB MA-CS 550 mg/Day (N=4) | DB Placebo (N=1) | OL MA-CS 550 mg/Day (N=0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspergillus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB MA-CS 550 mg/Day (N=4) | DB Placebo (N=1) | OL MA-CS 550 mg/Day (N=0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other